CLINICAL TRIAL: NCT03511209
Title: The Efficacy of Masked Tapering on Discontinuation of Hypnotics in Older Veterans
Brief Title: Discontinuation of Hypnotics in Older Veterans
Acronym: SWITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 17-234
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Insomnia
Keywords: Sleep Initiation and Maintenance Disorders; Hypnotics and Sedatives
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Only the participants and the outcome assessors will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBTI plus Taper method A (Experimental): Participants in this arm will receive Cognitive Behavioral Therapy for Insomnia (CBTI) plus the novel hypnotic tapering method.
  Interventions: Behavioral: CBTI plus taper method A
- CBTI plus Taper method B (Active Comparator): Participants in this arm will receive Cognitive Behavioral Therapy for Insomnia (CBTI) plus the usual tapering method used by the VA.
  Interventions: Behavioral: CBTI plus taper method B

INTERVENTIONS:
Behavioral: CBTI plus taper method A — This intervention includes CBTI plus the novel hypnotic tapering method.
  Arms: CBTI plus Taper method A
Behavioral: CBTI plus taper method B — This intervention includes CBTI plus the usual hypnotic tapering method used by the VA.
  Arms: CBTI plus Taper method B

SUMMARY:
Sleeping medications, called hypnotics, are often prescribed for insomnia. About one-quarter of Veterans use hypnotics (or bedtime alcohol). Older patients who use hypnotics fall more often and have worse memory than those who do not use them. Stopping hypnotics often reverses these problems. The Department of Veterans Affairs (VA) is trying to reduce hypnotic use among older adults. Currently, there are two main treatments to help patients stop using hypnotics. The first treatment involves a slow decrease in the daily dose until the hypnotic is ultimately discontinued. For safety, the process of decreasing the daily dose is usually supervised by a physician. The second is a treatment for insomnia called cognitive behavioral therapy for insomnia (CBTI).

This study will compare a novel hypnotic tapering method to the usual tapering method offered to older Veterans. The purpose of the study is to determine if the novel tapering method is more effective than the usual tapering method, both in terms of hypnotic discontinuation and improvement in insomnia severity.

Participants will be recruited from among Veterans 55 years and older who receive care from one VA Healthcare System. Following a baseline assessment, participants will be randomly assigned to one of the two 8-week treatment groups (66 participants per group). Each treatment group will receive CBTI, however, one group will receive the novel tapering program and the other group the usual tapering program. Follow-up assessments will be conducted at post-treatment and at 6-months after completion of the treatment.

If the novel tapering program is effective, it will represent a treatment option that can be offered to older Veterans who want to discontinue hypnotics. This tapering program could help VA healthcare providers adhere to clinical guidelines that recommend benzodiazepine discontinuation among older adults. A reduction in chronic hypnotic use may in turn reduce the risk of falls and hip fractures, which ultimately may improve the health and quality of life of older Veterans who receive healthcare at the VA.

DETAILED DESCRIPTION:
Hypnotics such as benzodiazepines and benzodiazepine receptor agonists are often prescribed for insomnia. Among Veterans attending outpatient clinics, approximately one-quarter use hypnotics (or bedtime alcohol). Hypnotics use is associated with an increased risk of falls and worse cognition in older adults. Discontinuing hypnotics often attenuates or reverses these negative effects, and the Department of Veterans Affairs (VA) has initiatives to reduce hypnotic use among older adults. Current discontinuation strategies focus on tapering off the hypnotic and/or treating insomnia symptoms. Common strategies include supervised gradual taper (SGT), cognitive behavioral therapy targeting hypnotic withdrawal (CBT-HW), cognitive behavioral therapy for insomnia (CBTI), and combination therapy (SGT+CBTI). Yet up to 40% of patients eventually resume use of hypnotics with these strategies, suggesting that other mechanisms need to be targeted to achieve and sustain high rates of non-use.

Objectives: 1) To assess the efficacy of a novel taper plus cognitive behavioral therapy-augmented program on hypnotic discontinuation among older Veterans, 2) to determine the impact of the the novel taper intervention on insomnia severity, 3) to assess the impact of the novel taper intervention on participants' beliefs and expectancies for using hypnotics to improve sleep quality and daytime function, and 4) to assess the efficacy of the novel taper intervention on balance and cognition.

To achieve these objectives, we propose to conduct a randomized clinical trial in older Veterans recruited from a single VA site. Veterans will undergo a 3-step screening process (letter with opt-out card, telephone screen, and in-person screen). Eligible participants (N = 132) will be randomized to 8 weeks of the novel taper intervention (CBTI+taper method A) or CBTI+taper method B. Follow-up assessments will be conducted at post-treatment and 6-months. Key 6-month outcomes will include hypnotic discontinuation and use (measured objectively through lab testing and medical record review/state prescription monitoring database query, and subjectively through sleep diary), insomnia severity, beliefs and expectations about hypnotics, balance, and cognition.

This hypnotic discontinuation program could be an important tool to help older Veterans who want to discontinue hypnotics to achieve this goal.

ELIGIBILITY:
Inclusion Criteria:

Age >= 55 years

* Use of lorazepam, alprazolam, temazepam, clonazepam, and/or zolpidem for current or prior insomnia symptoms 2 or more nights per week for at least 3 months
* Current or prior insomnia symptoms
* Available to attend weekly in-person or video sessions over 9 weeks

Exclusion Criteria:

High risk for complications in outpatient hypnotic discontinuation program:

* Seizure disorder
* Supratherapeutic/high baseline hypnotic dose (> diazepam-equivalent of 8 mg/night). Note that for individuals on > 1 of the targeted hypnotics, total baseline dose in diazepam-equivalents will be calculated & if > 8 mg/night, individual will be excluded.
* High risk of complicated withdrawal; benzodiazepine intoxication or current or past symptoms of complicated benzodiazepine/alcohol withdrawal (e.g., seizure, delirium at baseline)
* Polydrug use (e.g., chronic high dose opioids)
* Unable to keep study medications in secure location
* Evidence of prescription fraud (e.g., multiple prescriptions for same drug filled at VA and non-VA pharmacies, diversion)

Discontinuation of hypnotic not appropriate:

* Study-targeted hypnotic used to treat another clinical condition (e.g., Rapid Eye Movement sleep behavior disorder)
* Not willing to begin hypnotic discontinuation program

Poor candidate for CBTI:

* Presence of bipolar disorder
* Cognitive impairment (e.g., Mini-Mental State Examination < 24)
* Sleep/wake difficulty is better explained by another sleep disorder such as restless legs syndrome, narcolepsy, insufficient sleep syndrome, or circadian rhythm sleep-wake disorders
* Untreated sleep-disordered breathing defined as:

Apnea-hypopnea index (AHI) > 30 AHI between 15 and 30 and daytime sleepiness (Epworth Sleepiness Scale > 10)

* Medically/psychiatrically unstable (e.g., recent major hospitalization or planned major surgery during the study; psychosis, suicidal, active alcohol/substance abuse based on history and medical records)
* Unstable housing situation

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance H Fung, MD MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fung CH, Martin JL, Alessi C, Dzierzewski JM, Cook IA, Moore A, Grinberg A, Zeidler M, Kierlin L. Hypnotic Discontinuation Using a Blinded (Masked) Tapering Approach: A Case Series. Front Psychiatry. 2019 Oct 24;10:717. doi: 10.3389/fpsyt.2019.00717. eCollection 2019. PMID 31708806
- [Result] McCarthy M, Mak S, Kaufmann CN, Lum HD, Fung CH. Care coordination needs for deprescribing benzodiazepines and benzodiazepine receptor agonists. Res Social Adm Pharm. 2022 Apr;18(4):2691-2694. doi: 10.1016/j.sapharm.2021.06.025. Epub 2021 Jul 1. PMID 34229951
- [Result] Gutierrez L, Ghadimi S, Krall A, Hampson E, Grinberg AM, Moore AA, Dzierzewski JM, Alessi C, Martin JL, Fung CH. Posttraumatic Stress Disorder Risk and Benzodiazepine Dependence in Older Veterans with Insomnia Symptoms. Clin Gerontol. 2022 Mar-Apr;45(2):414-418. doi: 10.1080/07317115.2021.1954123. Epub 2021 Aug 4. PMID 34346855
- [Result] Ghadimi S, Grinberg A, Mitchell MN, Alessi C, Moore AA, Martin JL, Dzierzewski JM, Kelly M, Badr MS, Guzman A, Smith JP, Zeidler M, Fung CH. Sleep characteristics and use of multiple benzodiazepine receptor agonists in older adults. J Am Geriatr Soc. 2023 Dec;71(12):3924-3927. doi: 10.1111/jgs.18528. Epub 2023 Aug 1. No abstract available. PMID 37526436
- [Result] Fung CH, Alessi C, Martin JL, Josephson K, Kierlin L, Dzierzewski JM, Moore AA, Badr MS, Zeidler M, Kelly M, Smith JP, Cook IA, Der-Mcleod E, Ghadimi S, Naeem S, Partch L, Guzman A, Grinberg A, Mitchell M. Masked Taper With Behavioral Intervention for Discontinuation of Benzodiazepine Receptor Agonists: A Randomized Clinical Trial. JAMA Intern Med. 2024 Dec 1;184(12):1448-1456. doi: 10.1001/jamainternmed.2024.5020. PMID 39374004

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Behavioral Therapy for Insomnia (CBTI) Plus Taper Method A: Participants in this arm will receive Cognitive Behavioral Therapy for Insomnia (CBTI) plus the novel hypnotic tapering method.
  CBTI plus taper method A: This intervention includes CBTI plus the novel hypnotic tapering method.
- Cognitive Behavioral Therapy for Insomnia (CBTI) Plus Taper Method B: Participants in this arm will receive Cognitive Behavioral Therapy for Insomnia (CBTI) plus the usual tapering method used by the VA.
  CBTI plus taper method B: This intervention includes CBTI plus the usual hypnotic tapering method used by the VA.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy for Insomnia (CBTI) Plus Taper Method A | Cognitive Behavioral Therapy for Insomnia (CBTI) Plus Taper Method B
Started | 66 | 66
Completed | 63 | 60
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- CBTI Plus Taper Method A: Participants in this arm will receive CBTI plus the novel hypnotic tapering method.
  CBTI plus taper method A: This intervention includes CBTI plus the novel hypnotic tapering method.
- CBTI Plus Taper Method B: Participants in this arm will receive CBTI plus the usual tapering method used by the VA.
  CBTI plus taper method B: This intervention includes CBTI plus the usual hypnotic tapering method used by the VA.
- Total: Total of all reporting groups
Arm/Group | CBTI Plus Taper Method A | CBTI Plus Taper Method B | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (8.6) | 70.1 (7.7) | 69.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 54 | 54 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 5 | 16
  Not Hispanic or Latino | 55 | 61 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 6 | 14
  White | 51 | 52 | 103
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 6 | 2 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66 | 66 | 132
Insomnia Severity Index scale [Mean (Standard Deviation); unit: units on a scale] — Total score ranges from 0 to 28, with higher scores indicating greater insomnia severity
  units on a scale | 14.1 (6.9) | 14.2 (5.8) | 14.2 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Rates of Hypnotic Discontinuation
Description: The percentage of participants who had stopped taking a benzodiazepine or z-drug at follow-up. This outcome was measured with 7-day self-reported medication logs.
Time Frame: 6 months after treatment ends (which is an average of 8 months from randomization)
Measure: Count of Participants; unit: Participants
Arm/Group | CBTI Plus Taper Method A | CBTI Plus Taper Method B
Number analyzed (Participants) | 63 | 60
Participants | 48 | 36
Statistical Analysis 1: Comparison: CBTI Plus Taper Method A vs CBTI Plus Taper Method B; Compared CBTI plus Taper method A to CBTI plus Taper method B; Test type: Superiority; p = 0.056, Regression, Logistic; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.98 to 4.64], Standard Error of Mean 0.85

2. Primary Outcome: Insomnia Severity Index Score
Description: Mean score on Insomnia Severity Index. This 7-item scale measures self-reported severity of insomnia symptoms.
  Total score ranges from 0 to 28, with higher scores indicating greater insomnia severity.
Time Frame: 6 months after treatment ends (which is an average of 8 months from randomization)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI Plus Taper Method A | CBTI Plus Taper Method B
Number analyzed (Participants) | 66 | 66
score on a scale | 14.11 (6.86) | 14.20 (5.79)
Statistical Analysis 1: Comparison: CBTI Plus Taper Method A vs CBTI Plus Taper Method B; Test type: Superiority; p = 0.405, Mixed Models Analysis; Interaction contrast of Treatment Group (CBTI plus Taper method A vs. CBTI plus Taper method B) by Time (6 Months vs. Baseline); Mean Difference (Net) = -1.06, 95% CI 2-sided [-3.57 to 1.44], Standard Error of Mean 1.27

ADVERSE EVENTS:
Time Frame: Adverse events were collected over approximately 8-months (date of randomization until 6-months after treatment).
Arm/Group | CBTI Plus Taper Method A | CBTI Plus Taper Method B
All-Cause Mortality (participants affected / at risk) | 1/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 3/66 | 0/66
Other Adverse Events (participants affected / at risk) | 5/66 | 4/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBTI Plus Taper Method A (N=66) | CBTI Plus Taper Method B (N=66)
Hospitalization for respiratory viral illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Death from COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBTI Plus Taper Method A (N=66) | CBTI Plus Taper Method B (N=66)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
COVID-19 infection requiring ED visit (Infections and infestations) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Knee pain with torn meniscus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
parasomnia prior to receiving study medication (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT03511209/Prot_SAP_000.pdf